CLINICAL TRIAL: NCT03307863
Title: Effect of Anti-epileptic Drugs on Etonogestrel-releasing Implant Pharmacokinetics in Women With Epilepsy
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: We suspended the study for budget issues. It might be resumed in the future.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carolina Sales Vieira, Associate Professor, MD, PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2.140.103
Record Dates: First submitted 2017-09-27; First posted 2017-10-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Contraception; Drug Interactions
Keywords: etonogestrel implant; anti-epileptic drugs; pharmacokinetics
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: It is a non-randomized clinical trial (controlled clinical trial)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbamazepine-Implant (Experimental): Women with epilepsy using carbamazepine for at least 3 months will have an etonogestrel-releasing implant inserted
  Interventions: Drug: Carbamazepine-Implant
- Topiramate-Implant (Experimental): Women with epilepsy using topiramate for at least 3 months will have an etonogestrel-releasing implant inserted
  Interventions: Drug: Topiramate-Implant
- Implant (Active Comparator): Women without epilepsy and not using an anti-epileptic drug will have an etonogestrel-releasing implant inserted
  Interventions: Drug: Implant

INTERVENTIONS:
Drug: Carbamazepine-Implant — Women with epilepsy using carbamazepine for at least 3 months will have an etonogestrel-releasing implant inserted
  Arms: Carbamazepine-Implant
Drug: Topiramate-Implant — Women with epilepsy using carbamazepine for at least 3 months will have an etonogestrel-releasing implant inserted
  Arms: Topiramate-Implant
Drug: Implant — Women without epilepsy and not using an anti-epileptic drug will have an etonogestrel-releasing implant inserted
  Arms: Implant

SUMMARY:
Data on the interaction between the etonogestrel (ENG) implant and antiepileptic drug (AED) regimen are scarce. We will evaluated the effect of 2 AED regimens (1 including carbamazepine and the other topiramate) on the pharmacokinetic (PK) parameters of an ENG-releasing implant in women with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* women 18- 45 years old;
* with regular menstrual cycles;
* with BMI between 18 and 29.9 (kg/m2);
* who has selected the ENG implant as a contraceptive method;
* Using a stable antiepileptic drug regimen including carbamazepine or topiramate for ate least 3 months (only for women with epilepsy).

Exclusion Criteria:

* use of short-acting hormonal contraceptives in the month prior to enrollment;
* use of depomedroxyprogesterone acetate in the 6 months prior to enrollment;
* women with conditions classified as category 3 and/or 4 for etonogestrel implant use according to the World Health Organization Medical Eligibility Criteria for contraceptive use;
* drug or alcohol addiction;
* use of other drugs metabolized by CYP3A4 30 days prior to enrollment;
* non adherence to antiepileptic drug regimen (only for women with epilepsy);
* illiteracy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of ENG in women with epilepsy (WWE) using carbamazepine | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for area under the curve evaluation of ENG (AUC, 0-24 weeks). The plasma ENG AUC will be compared to that of women without epilepsy and without carbamazepine use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Plasma maximum concentration (Cmax) of ENG in women with epilepsy (WWE) using carbamazepine | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for evaluation of plasma Cmax of ENG. The plasma ENG Cmax will be compared to that of women without epilepsy and without carbamazepine use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Plasma minimum concentration (Cmin) of ENG in women with epilepsy (WWE) using carbamazepine | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for evaluation of plasma Cmin of ENG. The plasma ENG Cmin will be compared to that of women without epilepsy and without carbamazepine use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Time to maximum concentration (Tmax) of ENG in women with epilepsy (WWE) using carbamazepine | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for evaluation of Tmax of ENG. The Tmax of ENG will be compared to that of women without epilepsy and without carbamazepine use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.

SECONDARY OUTCOMES:
Bleeding pattern associated with etonogestrel implant use | Daily for 24 weeks
  Bleeding pattern (frequency, duration and number of bleeding/spotting days) associated with etonogestrel implant use will be evaluated in WWE using carbamazepine or topiramate and in women without epilepsy and without antiepileptic drug use
Area under the plasma concentration versus time curve (AUC) of ENG in women with epilepsy (WWE) using topiramate | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for area under the curve evaluation of ENG (AUC, 0-24 weeks). The plasma ENG AUC will be compared to that of women without epilepsy and without topiramate use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Plasma maximum concentration (Cmax) of ENG in women with epilepsy (WWE) using topiramate | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for evaluation of plasma Cmax of ENG. The plasma ENG Cmax will be compared to that of women without epilepsy and without topiramate use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Plasma minimum concentration (Cmin) of ENG in women with epilepsy (WWE) using topiramate | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for evaluation of plasma Cmin of ENG. The plasma ENG Cmin will be compared to that of women without epilepsy and without topiramate use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Time to maximum concentration (Tmax) of ENG in women with epilepsy (WWE) using topiramate | Prior to etonogestrel implant insertion and each 15 days for 24 weeks after implant placement
  Blood will be collected prior to ENG implant insertion and each 15 days for 24 weeks after implant placement for evaluation of Tmax of ENG. The Tmax of ENG will be compared to that of women without epilepsy and without topiramate use prior to ENG implant insertion and each 15 days for 24 weeks after implant placement.
Area under the plasma concentration versus time curve (AUC) of carbamazepine in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate AUC (0-8 hours) of carbamazepine
Plasma maximum concentration (Cmax) of carbamazepine in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate Cmax of carbamazepine
Plasma minimum concentration (Cmin) of carbamazepine in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate Cmin of carbamazepine
Time to maximum concentration (Tmax) of carbamazepine in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate Tmax of carbamazepine
Area under the plasma concentration versus time curve (AUC) of topiramate in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate AUC (0-8 hours) of topiramate
Plasma maximum concentration (Cmax) of topiramate in women with epilepsy (WWE) | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate Cmax of topiramate
Plasma minimum concentration (Cmin) of topiramate in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate Cmin of topiramate
Time to maximum concentration (Tmax) of topiramate in women with epilepsy (WWE) before and after ENG implant placement | Prior to implant placement and at 24 weeks of implant use
  Blood will be collected prior to etonogestrel implant use and at 24 weeks of its placement to evaluate Tmax of topiramate

OTHER OUTCOMES:
Acceptability | At 24 weeks of implant placement
  A questionnaire will be used to measure acceptability to etonogestrel implant by WWE
Satisfaction | At 24 weeks of implant placement
  A questionnaire will be applied to measure satisfaction of WWE with etonogestrel implant

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil